CLINICAL TRIAL: NCT04502745
Title: A Pilot Study of Endoscope-assisted, Minimally-invasive Cortical Access System (MICAS) for Chronic Subdural Evacuation
Brief Title: A Study to Evaluate Endoscope-assisted, Minimally-invasive Cortical Access System for Chronic Subdural Evacuation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of the flexible endoscope.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jamie J. Van Gompel, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20-005086
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): During clinically indicated surgery for subdural hematoma, the patient will undergo a single burr hole evacuation with the MICAS device with endoscopic assistance.
  Interventions: Device: Minimally Invasive Cortical Access System (MICAS)

INTERVENTIONS:
Device: Minimally Invasive Cortical Access System (MICAS) — Temporary surgical tool that provides access to the sub-dural space through the cranium.

SUMMARY:
The purpose of this study is to evaluate a less-invasive alternative to the currently available method of removing aging blood in the subdural space.

ELIGIBILITY:
Inclusion Criteria:

* Must be 55 years of age or greater.
* Have a clinically symptomatic chronic subdural hematoma greater than 1 cm in maximal thickness and be judged clinically to need subdural evacuation.

Exclusion Criteria:

* Failure to obtain consent.
* Vulnerable study population.
* Any need for chronic anticoagulation.
* Pregnancy (verified by pregnancy testing at screening or medical history of a hysterectomy, oophorectomy, or post-menopausal).Prior surgery for subdural hematoma.
* Glasgow Coma Scale (GCS) less than 8.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Incidence of all serious adverse events | 3 years
  Number of adverse events including unanticipated adverse device effects

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Van Gompel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials